CLINICAL TRIAL: NCT05271110
Title: A Population-based Assessment of Curative Intended Multimodal Treatment in Patients With Oligometastatic Pancreatic Cancer, Responsive to Neoadjuvant Chemotherapy - ScanPan 1 - A Scandinavian Prospective Multicenter Study
Brief Title: Surgery for Liver Metastases From PDAC
Acronym: ScanPan1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Lund University (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Umeå (Other); University of Southern Denmark (Other); University of Copenhagen (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bergthor Björnsson, Associate Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScanPan 1
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Disseminated Pancreatic Cancer
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: A prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment cohort (Experimental): Adult patients (ECOG 0-1) with a resectable (or previously resected) PDAC and either synchronous or metachronous liver metastases are the target population of this study.
  Interventions: Procedure: Liver resection (ablation)

INTERVENTIONS:
Procedure: Liver resection (ablation) — Treatment of liver metastases from pancreatic cancer by surgery or ablation

SUMMARY:
Dissemination from pancreatic ductal adenocarcinoma (PDAC) occurs in clinical practice either in the form of recurrence after initial treatment with curative intent resection (metachronous) or more frequently prevails already at the time of diagnosis (synchronous). Traditionally, metastatic pancreatic cancer (mPDAC) is considered not to be eligible for meaningful aggressive therapies to be implemented. However, with the development of local as well as more effective systemic therapeutic regimens a variety of clinical situations have to be reevaluated. For instance, recent reports have indicated an option for maintained or even prolonged survival after resections and/or ablations of oligometastatic pancreatic cancer (OMDPDAC), as represented by a single or few liver metastasis (es). These reports are burdened by methodological weaknesses such as being retrospective, single institution and reporting only from highly selected case series.

A common denominator of acceptable outcome is, however, that all metastatic lesions have been preoperatively treated and responded to chemotherapy, indicating an advantageous tumor biology.

Hence an unbiased approach, including neo-adjuvant chemotherapy before any aggressive local treatment must be explored to the updated management opportunities in terms of assessing the prevalence, safety, feasibility, tolerability and possible disease control options.

Primary objective (clinical): To prospectively investigate (on an intention to treat basis) the safety, feasibility, tolerability and clinical outcomes of all patients with PDAC presenting with limited metastatic disease, where a treatment option can be launched with the ambition of local disease control and eventually better survival.

The cohorts to be included are:

Primary cohort: Patients with liver limited (metachronous and synchronous) metastasis(es) due to PDAC. This cohort is further subdivided to:

Limited liver disease. Extended liver disease. Secondary cohort: Patients with OMDPDAC and at least one extrahepatic manifestation of PDAC.

Secondary objective (translational) is to improve the understanding of PDAC liver metastases biology by studying the mechanistic aspects of metastases invasion as well as intra- and peri-tumoral liver metastatic niche, and by charting the cellular composition of liver metastases on single cell level with a focus on the impact of cellular interactions on tumor cell growth and differentiation. Furthermore, the study aims to identify blood-based biomarkers of response to oncologic/surgical treatment.

DETAILED DESCRIPTION:
Dissemination from pancreatic ductal adenocarcinoma (PDAC) occurs in clinical practice either in the form of recurrence after initial treatment with curative intent or more frequently is manifested already at the time of diagnosis. Traditionally corresponding disease states are considered not to be eligible for meaningful aggressive therapies to be implemented. Instead, palliative therapies are instituted with a very limited survival. However, with the development of local as well as more effective systemic therapeutic regimens, a variety of clinical situations must be reevaluated.

In PDAC, disseminated to the liver, the traditional view as that the corresponding lesions are non-treatable by aggressive chemotherapy followed by surgical interventions and generally, surgery has been considered obsolete in this patient cohort5. Despite these early discouraging results there are some reports, from selected cohorts, indicating more promising survival rates after resection of metastasis(es) than ever earlier described6. Moreover, during recent years there has been significant improvement in the efficacy of chemotherapy regimens available for patients with localized as well as disseminated PDAC that may enhance the effect of surgical removal of macroscopic tumor manifestations.

The same may be true for alternative limited manifestations of metastatic PDAC disease. Hence an unbiased approach must be explored to the updated management opportunities in terms of assessing the incidence, safety, feasibility, tolerability and possible disease control options.

According to the Swedish and Danish pancreatic cancer registry the overall median survival (OS) of patients with pancreatic cancer is about 6-7 months while studies demonstrate 9-15 months median survival when palliative chemotherapy is used7, 8.

Hitherto, no prospective, population-based study, with intention to treat design, has been presented to define the role of aggressive oncological regimens with successive macroscopic eradication of tumor lesions as exemplified by surgery in disseminated PDAC. The evidence at hand comes from retrospectively collected and selected cohorts where comparison is often made to surgical palliation alone (intestinal bypass surgery) or best supportive care. The reported median survival after surgery varies widely from 7.6 months to as long as 56 months9. A recent case matched study suggested that in selected cases, surgery may improve median survival from about 1 to 2 years10. Corresponding data just reflect the large impact of selection on either the intervention and/or the control group. The main drawback of the available literature is the general lack of population based, intention to treat data and lack of clear definition of disease stages that severely limit the usefulness of these results in clinical decision making.

The evidence for applying invasive treatment for extrahepatic dissemination of PDAC is even more limited although dissemination to the lungs may be associated with somewhat longer overall survival than other locations 11.

Despite increasing evidence for some role of updated multimodal treatment options in disseminated PDAC there is a strong need for an intention to treat designed prospective, population-based study to investigate the value of corresponding regimens in PDAC.

Eligible for enrolment are all patients presenting with the following characteristics:

Primary cohort; Synchronous or metachronous liver metastasis(es) from PDAC without signs of extra hepatic disease. This cohort is subdivided:

* Limited liver disease: Synchronous or metachronous uni- or bilobar liver metastasis(es) from PDAC. The number of metastases shall be < 4 and the largest < 5 cm (2 cm if ablative treatment is planned) and no signs of extrahepatic dissemination. This cohort forms the basis for sample size calculation and primary outcome.
* Extended liver disease: Liver limited metastasis that do not fit into the limited liver disease cohort but are still evaluated at a multidisciplinary conference and judged as amendable for treatment with curative intent Secondary cohort; PDAC patients with limited (unilocular) dissemination to intra- or extra-abdominal locations rendering the lesion(s) amenable to either; SBRT, alternative external radiation options, surgery, thermal ablation or a combination of these. Patients with loco-regional recurrences of PDCA as defined as those detected in the remaining part of the resected organs (e.g. the gastric or pancreatic remnant), in the anastomotic area, the anatomic area representing the original resection bed, regional remaining lymph nodes. Patients with isolated loco-regional recurrences as defined as those emerging and detected in the above-mentioned sites, and with no signs of distant metastases.

All these patients are identified at multidisciplinary tumor boards in each participating center.

Patients deemed fit for oncological treatment are enrolled and chemotherapy started. After at least 2 months of chemotherapy patient status is reevaluated with CT scan/MRI and PET-CT and in case of response (stable disease or regression according to the RECIST 1.1 criteria) and also evaluating tumour markers (CA19.9), local treatment is given.

For inclusion in the Primary "Limited liver disease" cohort" a minimum of 4 months chemotherapy treatment is given.

If response is not achieved on initial oncological treatment, further treatment may be given and disease status re-evaluated every other month as long as considered clinically relevant-meaningful. Patients that do not achieve stable disease/regression will continue palliative treatment as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

Confirmed PDAC with synchronous or metachronous dissemination isolated in the liver (primary cohort) or other dissemination as described in chapter 7.1. where the local tumour board find indication for curative treatment attempt.

The confirmation of PDAC before chemotherapy is not regulated by the protocol but EUS guided biopsies directed to the primary tumour or a site of recurrence/dissemination is recommended whereas a percutaneous approach towards liver lesion(s) can be an alternative diagnostic approach; radiology and elevated serum tumor markers may guide diagnosis in exceptional cases, for which, e.g., pathological sampling fails.

Metastases are defined as synchronous when liver tumors are detected simultaneously with the primary tumor or within the first 6 months thereafter. All other tumors are regarded as metachronous metastases or locally recurrent disease (when applicable).

The same definition applies to localized lesions detected intra- as well as extra-abdominally.

Patients treated due to the radiological appearance and or elevated CA-19.9 levels despite negative biopsies are accepted for inclusion into the study

To be included in "Limited liver desease":

Up to 4 liver metastases treatable with liver resections (without volume expansion of the future liver remnant)/thermal ablations/RFA/IRE (largest diameter < 5 cm and for ablative techniques < 2 cm).

Age 18 years or older ECOG 0-1 Any resectable (including borderline resectable, but without need for arterial reconstruction) (before or after neoadjuvant treatment) PDAC Patient can understand verbal and written information

Exclusion Criteria:

Age less than 18 years ECOG >2 Patient is not able to understand the verbal and written information Progression of tumor (RECIST 1.1) during or after chemotherapy Distant metastases outside the liver (applies only to the primary cohort) Other malignancy within 2 years, the prognosis of which may affect the evaluation of the therapeutic outcome.

Major non-pancreatic surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery Uncontrolled (bacterial or fungal) infections Significant concomitant diseases preventing the safe administration of study drugs or likely to interfere with study assessments Uncontrolled angina pectoris; cardiac failure or clinically significant arrhythmias Continuous use of immunosuppressive agents (Corticoids are allowed) Neuropathy >grade 1 (CTCAE, v 5.0) Pregnancy or breast feeding Patients (M/F) with reproductive potential not implementing adequate contraceptive measures Pre-defined need for arterial reconstruction to resect primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of surgery | Up to 90 days after surgery
  Safety of liver metastases treatment with surgery or ablation as measured by the proportion of patients experiencing severe complications (defined by the Clavien-Dindo classification)
Feasibility of treatment | 3 years
  Measured as the proportion of patients starting neoadjuvant chemotherapy that finally get invasive treatment for their liver metastases

SECONDARY OUTCOMES:
Chemotherapy associated morbidity | 3 years
  Measured as the number of adverse events occuring during neoadjuvant chemotherapy
Surgical morbidity according to the Clavien-Dindo classification | 90 days after surgery
  Classified according to the Clavien-Dindo classification and reported as the most severe complication
Surgical morbidity according to the CCI (comprehensive complication index) | 90 days post operatively
  All complications occuring up to 90 days after surgery are combined in a CCI for each patient
Pos operative pancreatic fistula (POPF) | 90 days post operatively
  Defined according to established criteria, proportion of patients experiencing POPF will be reported
Post pancreatectomy hemorrhage (PPH) | 90 days post operatively
  Defined according to established criteria, proportion of patients experiencing PPH will be reported
Delayed gastric emptying (DGE) | 90 days post operatively
  Defined according to established criteria, proportion of patients experiencing DGE will be reported
R0 resection rate of liver metastasis | 3 yeras
  Defined as <1mm margin on pathology assessment
Histological tumor response | 3 years
  Graded on pathology assessment as the proportion of viable tumour cells in the specimen
Overall survival | 5 years
  Calculated with the Kaplan-Meier method 2 years after last surgery
Progression free survival | 5 years
  Calculated with the Kaplan-Meier method 2 years after last surgery
Disease free survival | 5 years
  Calculated with the Kaplan-Meier method 2 years after last surgery
Quality of life after surgery | 5 years
  Measured with EQ5D before and up to 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Linkoping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasselgren K, Williamsson C, Wennerblom J, Ghorbani P, Liljefors MG, Huhta H, Heby M, Mansson C, Johansson MI, Elander NO, Nortunen M, Kallio R, Halimi A, Ohlund D, Sandstrom P, Sparrelid E, Bjornsson B. Prospective evaluation of surgical treatment of liver metastasizing pancreatic cancer - ScanPan study protocol. BMC Surg. 2025 Jul 19;25(1):299. doi: 10.1186/s12893-025-02983-w. PMID 40682051